CLINICAL TRIAL: NCT01690013
Title: Life Quality and Health in Patients With Klinefelter Syndrome - a Questionnaire Survey
Brief Title: Life Quality and Health in Patients With Klinefelter Syndrome
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-41-0666
Record Dates: First submitted 2012-09-11; First posted 2012-09-21 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2012-09

CONDITIONS: Klinefelter Syndrome; Quality of Life; Physical Disorders; Mental Disorders
MeSH Terms: conditions — Klinefelter Syndrome; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Klinefelter: Men with Klinefelter syndrome
- Control: Men from the general population, matched by age, education and zipcode.

SUMMARY:
Klinefelter syndrome is the most common sex-chromosome disorder in men with a prevalence of 1 in 660 men. The syndrome is associated with hypogonadism. Many patients with Klinefelter syndrome have psychological complaints and physical discomfort. Some patients report a positive effect of testosterone treatment, whereas others do not.

The aim of this study is:

(i) To investigate quality of life in patients with Klinefelter syndrome. (ii) To investigate functional, physical and mental health in patients with Klinefelter syndrome.

Questionnaire concerning mental and physical health and life quality are sent out to patients with KS and to age-, educational- and zipcode-matched men from the general population. The questionnaire include questions about housing, income, marital status, fatherhood, medication, chronic disease,school and education, attachment to the labor, sexual and erectile function, life quality, mental and physical health, satisfaction with life and symptoms of attention deficits hyperactivity disorders.

ELIGIBILITY:
For the Klinefelter group:

Inclusion Criteria:

* Verified Klinefelter syndrome

Exclusion Criteria:

* none

For the control group:

Inclusion Criteria:

* age-,educational,and residence-matched

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Klinefelter patients is recruited from endocrinology, genetics and fertility clinics in Denmark.
  An age-, educational, and zipcode-matched control group was created from Statistics Denmark by extracting five randomly selected men for each KS subject
Sampling Method: Non-Probability Sample
Enrollment: 452 (Actual)
Dates: Start 2012-09; Primary Completion 2013-01 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Quality of life | 3 month
  Quality of life score is measured with the WHOQOL-Brief questionnaire
Satisfaction with life | 3 month
  Satisfaction with life is measured with the SWLS - Satisfaction with Life Scale
ADHD symptoms | 3 month
  ADHD symptoms are measured by Adult ADHD Self-Report Scale (ASRS-v1.1) Symptom Checklist
General health | 3 month
  General health is measured by SF-36 questionnaire
Erectile function | 3 month
  Erectile function is measured by the International index of erectile function (IIEF-5) as a diagnostic tool for erectile function.

OTHER OUTCOMES:
Housing | 3 month
Fatherhood | 3 month
School and educational | 3 month
  Information about school and education
Income | 3 month
Attachment to the labor | 3 month
  working position, working hour, period of sick leave
Marital status | 3 month
Medication | 3 month
Chronic disease | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Claus H Gravholt, MD, Dr.med., Principal Investigator — Medical Department M, Aarhus Universityhospital, Aarhus
Locations (1):
- Medical Department M, Aarhus Universityhospital, Aarhus, Denmark